CLINICAL TRIAL: NCT04355845
Title: A PHASE 1, FIXED-SEQUENCE, OPEN LABEL STUDY TO EVALUATE THE EFFECT OF PF-06651600 ON PHARMACOKINETICS OF SINGLE DOSE SUMATRIPTAN IN HEALTHY PARTICIPANTS
Brief Title: A STUDY TO EVALUATE THE EFFECT OF PF-06651600 ON PHARMACOKINETICS OF SINGLE DOSE SUMATRIPTAN IN HEALTHY PARTICIPANTS.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B7981025
Record Dates: First submitted 2020-04-06; First posted 2020-04-21 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
Keywords: PF-06651600; Sumatriptan; Drug-drug interaction study; Pharmacokinetics
MeSH Terms: interventions — Sumatriptan; PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sumatriptan and PF-06651600 DDI (Experimental): In Period 1, participants will receive a single oral 25 mg dose of sumatriptan on Day 1 in the morning. In Period 2 on Day 1, participants will receive a single oral 25 mg dose of sumatriptan and a single 400 mg oral dose of PF-06651600 in the morning. In Period 3 participants will receive a single 400 mg oral dose of PF-06651600 in the evening of Day 1, and then a single oral 25 mg dose of sumatriptan in the morning of Day 2.
  Interventions: Drug: Sumatriptan; Drug: PF-06651600

INTERVENTIONS:
Drug: Sumatriptan — 25 milligrams (mg) single dose tablet
Drug: PF-06651600 — PF-06651600 400 mg single dose

SUMMARY:
Study to evaluate the effect of pf-06651600 on pharmacokinetics of single dose sumatriptan.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female participants who are healthy as determined by medical evaluation including medical history, full physical examination which includes BP and pulse rate measurements, clinical laboratory tests, and 12-lead ECG.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), diabetes or of the contraindications as per the USPI for IMITREX.
* 10-year risk of atherosclerotic cardiovascular disease (based on ASCVD Risk Estimator) ≥7.5%.
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Systemic therapy with any of the medications that are MAO-A inhibitors within 14 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. Concomitant use of any ergotamine-containing or ergot-type medication (like dihydroergotamine or methysergide), or other 5-HT agonist (Section 6.5) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* Known participation in a clinical trial of PF-06651600 within 60 days prior to the first dose of investigational product; participation in any clinical trial of PF-06651600 and the participant experienced AE that led to discontinuation or had an SAE that in the judgment of the investigator were PF-06651600-related.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Sumatriptan area under the curve (AUC) extrapolated to infinite time. | Predose, at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post sumatriptan dose.
Sumatriptan (Cmax) maximum plasma concentration | Predose, at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post sumatriptan dose.
Sumatriptan AUC last PK sample. | Predose, at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post sumatriptan dose.

SECONDARY OUTCOMES:
Number of participants with significant changes from baseline in vital signs. | Baseline through Period 3 Day 4 (Day 8).
Number of participants with significant changes from baseline in electrocardiogram (ECG). | Baseline through Period 3 Day 4 (Day 8).
Number of participants with significant changes from baseline in lab tests. | Baseline through Period 3 Day 4 (Day 8).
Number of participants with adverse events. | Baseline through to Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981025